CLINICAL TRIAL: NCT01963520
Title: Prospective Study of Patients Treated for Prosthetic Hip Infection and Followed for at Least 2 Years
Brief Title: Prosthetic Hip Infections: Prospective Study
Acronym: PHIPS
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, Dr Valerie ZELLER, Investigator coordinator, Groupe Hospitalier Diaconesses Croix Saint-Simon
Other Study IDs: GHDCSS-01
Record Dates: First submitted 2013-09-26; First posted 2013-10-16 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Hip Prosthesis Infection
Keywords: Hip prosthesis infection; Reinfection; Excision-synovectomy; One stage/two stage revision; Antibiotherapy
MeSH Terms: conditions — Reinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Data from large prospective cohort studies of prosthetic joint infections are lacking.

Aim of this study: analyzing prospectively the incidence of reinfection in patients with prosthetic hip infections who underwent surgery and received antibiotic therapy.

Hypothesis: to confirm in a large group that the incidence of reinfection after excision -synovectomy in acute prosthesis hip infection is 30% and 15% for chronic infection after exchange arthroplasty (one or two stage exchange).

DETAILED DESCRIPTION:
Aim of the study: to analyze the incidence of reinfection in patients with prosthetic hip infection who underwent surgery and received antibiotic therapy Methods: prospective cohort study in a French referral center for osteoarticular infections from November 2002 to March 2010. Population

* all patients who consented to participate in the study with prosthetic hip infections treated by:
* debridement-synovectomy for acute infection or with one-stage or two-stage
* exchange arthroplasty or resection arthroplasty for chronic infection
* antibiotic therapy

Outcome:

* Follow-up: minimum of 2 years
* Events monitored: reinfection including relapse and new infection, joint revision for mechanical reasons, prosthetic hip infection related and non-related deaths

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip arthroplasty infection
* Surgical treatment: either debridement-synovectomy and prosthesis retention for acute infection or one or two-stage exchange arthroplasty or resection arthroplasty for chronic infection
* Antibiotic therapy
* Signed informed consent

Exclusion Criteria:

* Prolonged suppressive antibiotic therapy
* No surgical treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hip arthroplasty infection who underwent surgery and received antibiotic therapy in a specialized French orthopaedic center for bone and joint infection.
Sampling Method: Non-Probability Sample
Enrollment: 347 (Actual)
Dates: Start 2002-08-02; Primary Completion 2010-03 (Actual); Study Completion 2015-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence of reinfection (relapse and new infection) | 2 years
  The aim of this study was to prospectively determine the incidence of reinfection in patients with prosthetic hip infection after two years of follow up.

SECONDARY OUTCOMES:
Incidence and causes of mechanical revision | 2 years
Incidence and causes of death: infection or treatment related death, unrelated death | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Valerie ZELLER, MD, Principal Investigator — Diaconesses Croix Saint-Simon Hospital Group, Paris, France
Locations (1):
- Diaconesses Croix Saint-Simon Hospital Group, Paris, France

REFERENCES:
- [Result] Tsukayama DT, Estrada R, Gustilo RB. Infection after total hip arthroplasty. A study of the treatment of one hundred and six infections. J Bone Joint Surg Am. 1996 Apr;78(4):512-23. doi: 10.2106/00004623-199604000-00005. PMID 8609130